CLINICAL TRIAL: NCT05447013
Title: Generation of SARS-CoV-2-specific T Lymphocytes From Recovered Donors and Administration to High-risk COVID-19 Patients
Acronym: CoV-2-STs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Papanicolaou Hospital (Other)
Collaborators: General Hospital Of Thessaloniki Ippokratio (Other)
Responsible Party: Principal Investigator, Evangelia Yannaki, PI, Director of the Gene and Cell Therapy Center, Hematology-HCT Unit, George Papanicolaou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoV-2-STs-001
Record Dates: First submitted 2022-06-30; First posted 2022-07-07 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Severe COVID-19
Keywords: COVID-19; Virus-specific T cells; SARS-CoV-2; Coronavirus-specific T cells; 2021-001022-22
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- For Phase II: Arm A (Experimental): Standard of care (SOC) and Coronavirus-specific T cells (CoV-2-STs)
  Interventions: Biological: Coronavirus-2-specific T cells
- For Phase II: Arm B (Active Comparator): Standard of care (SOC)
  Interventions: Other: standard of care (SOC)

INTERVENTIONS:
Biological: Coronavirus-2-specific T cells — Coronavirus-2-specific T cells ex vivo expanded from selected COVID-19 recovered donors
  Arms: For Phase II: Arm A
Other: standard of care (SOC) — standard of care (SOC)
  Arms: For Phase II: Arm B

SUMMARY:
Open-label phase I (single-center)/ phase II (multicenter) with randomization 2:1

DETAILED DESCRIPTION:
Phase I (single-center): The investigators will administer CoV-2-STs in a dose escalation regimen of 2 dose levels (DL1: 1,5x10^7 CoV-2-STs in total; DL2: 2x10^7 CoV-2-STs/m^2). 3 patients will be treated at each dose level (traditional 3+3 design) following by a 12-day wait period to assess safety of the infusions prior to escalating the next dose level (maximum 12 patients). The maximum tolerated dose will be determined Phase II (multicenter): Randomization 2:1, 60 patients will receive the standard of care (SOC) plus CoV-2-STs (ARM A) at the optimum dose which will be determined in phase I and 30 patients will receive only SOC (Arm Β) Phase II (multicenter, extension): Randomization 2:1, 53 patients will be enrolled in Arm A to receive SOC and up to two doses of COV-2-STs and 27 patients will receive only SOC.

Randomization: Patients who meet the eligibility criteria after signing the informed consent form they will randomly be assigned at 2:1 ratio to each of the 2 treatment groups. Patients assigned to arm A will be HLA-typed for HLA-A, B and DRB1 within 24h, and a suitable for them T cell product will be selected from the cell bank. If a suitable product is found, they will continue to arm A, otherwise, they will be assigned to arm B.

Objectives:

i) To determine the feasibility of establishing a bank with GMP-compliant generated SARS-CoV-2 specific T-cells (CoV-2-STs), well-characterized in terms of specificity, phenotype and expression of human leucocyte antigens (HLA), which will be produced by 30 COVID-19 recovered donors with broad HLA diversity in order to be suitable for administration to at least 90 COVID-19 patients ii) To determine the safety of CoV-2-ST administration as cellular immunotherapy in COVID-19 patients, who meet specific inclusion criteria iii) To determine the efficacy of CoV-2-ST administration as cellular immunotherapy in COVID-19 patients, who meet specific inclusion criteria

ELIGIBILITY:
Inclusion Criteria: Hospitalized patients, SARS-CoV-2 PCR positive, within 8 days from the onset of the symptoms (immunosuppressed patients are excluded from the time limit when they become chronic carriers of the virus), who have:

* Pneumonia or/and SatO2 ≤94% on room air or/and respiratory rate ≥24breaths/min AND
* lymphopenia CD3+≤650/μl or/and ALC≤1000/microl AND
* Increased values of D-dimers (≥2Χ) or/and ferritin (>1000ng/ml) or/and CRP (≥3Χ) or/and LDH (≥2Χ)

Exclusion Criteria:

* Age ≤18 and ≥80 years old
* Onset of symptoms >8 days (immunosuppressed patients are excluded from the time limit when they become chronic carriers of the virus)
* Corticosteroid administration at a dose of >0.75mg/kg (methylprednisolone equivalent)
* Multiple organ failure
* ARDS (acute respiratory distress syndrome)
* Mechanical ventilation
* Patients who received ATG, or Campath, or other T-cell-suppressing monoclonal antibody within 28 days prior to admission
* Patients with concomitant confirmed infection from another pathogen or with very high procalcitonin (PCT) that may indicate additional infection
* Enrollment in another clinical trial
* Pregnancy
* Inability to sign informed consent form
* Judged ineligible by at the treating physician (treating physician's discretion)
* Bilirubin ≥2x of upper normal limit
* AST ≥ 2x of upper normal limit
* Creatinine ≥ 2x of upper normal limit or with dialysis/hemodialysis needs
* Karnofsky score ≤50

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of a CoV-2-STs bank | Within 2 months before recruitment initiation
  • Thirty, multi-dose, GMP-generated and released CoV-2-ST products
Establishment of a CoV-2-STs bank of broad HLA coverage | Within 2 months before recruitment initiation
  CoV-2-ST products of a broad HLA repertoire
Pharmacodynamic endpoint-1 (Phase I) | Up to the completion of Ph I
  •Determination of optimal dose (maximum tolerated dose)
Pharmacodynamic endpoint-2 (Phase I and II) | Up to the completion of Ph I and II
  • In vivo expansion of CoV-2-STs after administration
Pharmacodynamic endpoint-3 (Phase II) | Up to the completion of Ph II
  • Persistence of circulating donor CoV-2-STs by microchimerism analysis
Efficacy endpoint-1 (Phase II) | Day 30 and Day 60 (end of follow up)
  • Recovery and time to recovery. Recovery is defined as a value of 1 to 3 on the 8-point WHO ordinal scale (OS). Time to recovery is the days passed from Day 0 to the 1st day of a score 1 to 3 on the OS for those who recovered or the days passed from Day 0 to the last follow-up for the rest.
Efficacy endpoint-2 (Phase II) | Day 30 and Day 60 (end of follow up)
  • Survival by days 30 and 60. Survival is defined as the time-to-event from Day 0 to the date of death or the last follow-up
Safety endpoints (Phase I and II) | End-of-follow up (day 60) for all patients in Ph I and Ph II
  * acute toxicity related to the CoV-2-ST infusion, by clinical and laboratory assessments
  * cytokine release syndrome, by clinical and laboratory assessments
  * number of adverse and/or serious adverse events

SECONDARY OUTCOMES:
Efficacy endpoint-1 (Phase II) | Day 30 for all enrolled patients
  -Clinical status by the 8-point WHO Ordinal Scale on day 30
Efficacy endpoint-2 (Phase II) | End-of-follow up (day 60)
  * time to improvement by 1 & 2 categories from day 0 according to the 8-point Ordinal Scale
  * time to PCR negativity
  * time to lymphopenia recovery
  * hospitalization time ( day 0 to discharge)
Efficacy endpoint-3 (Phase II) | Day 20 for all enrolled patients
  Percentage of patients with negative PCR by day 20
Safety endpoint (Phase I and II) | End-of-follow up (day 60)
  •Graft versus host disease (GvHD), by clinical and laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Yannaki, MD,PI, Principal Investigator — George Papanicolaou Hospital
Locations (2):
- Greece (2):
  - General Hospital of Thessaloniki Ippokratio- 2nd Propedeutic Department of Internal Medicine, Thessaloniki
  - George Papanikolaou Hospital - Gene and Cell Therapy Center- Hematology Dpt- Hematopoietic Stem Cell Transplant Center, Thessaloniki

IPD SHARING:
Plan to Share IPD: No